CLINICAL TRIAL: NCT02222870
Title: Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Quadrivalent, Influenza Vaccine (2014-2015 Formulation)
Brief Title: Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Quadrivalent, Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC56; U1111-1143-8966 (Other: WHO)
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Quadrivalent Influenza Virus Vaccine (No Preservative); Fluzone®
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone Study Group 1 (Experimental): Participants at 6 months to < 36 months age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative
- Fluzone Study Group 2 (Experimental): Participants at 3 years to < 9 years of age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative

INTERVENTIONS:
Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative — 0.25 mL, Intramuscular (Pediatric Dose, 2014-2015 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Fluzone Study Group 1
Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular (2014-2015 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Fluzone Study Group 2

SUMMARY:
The study will evaluate the safety and immunogenicity of the 2014-2015 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule, in accordance with the Advisory Committee on Immunization Practices (ACIP) recommendations, in children 6 months to < 9 years of age.

Objective:

* To describe the safety of the 2014-2015 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule, in accordance with ACIP recommendations, in children 6 months to < 9 years of age.

Observational objectives:

* To describe the immunogenicity of the 2014-2015 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule in accordance with ACIP recommendations, in children 6 months to < 9 years of age.
* To submit available sera from each subject to Center for Biologics Evaluation and Research (CBER) for further analysis by the WHO, the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
Participants will be assigned to the appropriate age group based on the age at the time of enrollment. Participants will receive a dose of Fluzone Quadrivalent vaccine, those for whom 2 doses of influenza vaccine are recommended per ACIP guidance, will receive a second dose during Visit 2 (28 days after Visit 1).

Solicited adverse event (AE) information will be collected for 7 days after each vaccination, unsolicited AE information will be collected from Visit 1 to Visit 2, or to Visit 3 for those subjects receiving 2 doses. Serious adverse event (SAE) information will be collected the study. Immunogenicity will be evaluated in all participants prior to vaccination and at Day 28 after the final vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 6 months to < 9 years of age on the day of first study vaccination (study product administration)
* Subject and parent/legally acceptable representative are willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Assent form has been signed and dated by subjects 7 to < 9 years of age, and informed consent form has been signed and dated by parent(s) or another legally acceptable representative for subjects 6 months to < 9 years of age.
* For subjects 6 months to < 12 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information).
* History of serious adverse reaction to any influenza vaccine.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2 for subjects receiving 1 dose of influenza vaccine or Visit 3 for subjects receiving 2 doses of influenza vaccine.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study.
* Prior vaccination with any formulation of 2014-2015 influenza vaccine.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré Syndrome.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Identified as a natural or adopted child of the Investigator or an employee with direct involvement in the proposed study.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Bardstown, Kentucky
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 19 August 2014 to 06 November 2014 at 2 clinical sites in the United States.
Pre-assignment Details: A total of 60 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated in the study.
Groups:
- 6 to < 36 Months of Age: Participants 6 to < 36 months of age who received 1 or 2 intramuscular dose(s) of Fluzone Quadrivalent vaccine.
- 3 to < 9 Years of Age: Participants 3 to < 9 years of age who received 1 or 2 intramuscular dose(s) of Fluzone Quadrivalent vaccine.
Period: Overall Study
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 25.0 (8.3) | 66.9 (21.8) | 45.9 (26.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Solicited Injection-site: 6 to < 36 months - Tenderness, Erythema, and Swelling; 3 to < 9 years - Pain, Erythema, and Swelling. Solicited systemic reactions: 6 to < 36 months - Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability; 3 to < 9 years - Fever, Headache, Malaise, and Myalgia.
  Grade 3: Fever, > 39.5˚C (6 to < 36 months), ≥ 39.0˚C (3 to < 9 years); Vomiting, ≥ 6 episodes/24 hours or requires parenteral hydration; Crying abnormal, > 3 hours; Drowsiness, Sleeping often/difficult to wake; Appetite lost, Refuses ≥ 3 or most meals; Irritability, Inconsolable; Headache, Malaise, and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-any injection
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Number analyzed (Participants) | 30 | 30
Percentage of participants
  Injection-site Tenderness (N=30, 0) | 70.0 | NA — Event was not assessed in this group
  Grade 3 Injection-site Tenderness (N=30, 0) | 3.3 | NA — Event was not assessed in this group
  Injection site Pain (N=0, 30) | NA — Event was not assessed in this group | 73.3
  Grade 3 Injection site Pain (N=0, 30) | NA — Event was not assessed in this group | 10.0
  Injection-site Erythema | 50.0 | 66.7
  Grade 3 Injection-site Erythema | 0.0 | 0.0
  Injection-site Swelling | 23.3 | 43.3
  Grade 3 Injection site Swelling (6 to <36 months) | 0.0 | 0.0
  Fever | 20.7 | 3.3
  Grade 3 Fever | 0.0 | 0.0
  Vomiting (N=30, 0) | 16.7 | NA — Event was not assessed in this group
  Grade 3 Vomiting (N=30, 0) | 0.0 | NA — Event was not assessed in this group
  Crying abnormal (N=30, 0) | 33.3 | NA — Event was not assessed in this group
  Grade 3 Crying abnormal (N=30, 0) | 0.0 | NA — Event was not assessed in this group
  Drowsiness (N=30, 0) | 30.0 | NA — Event was not assessed in this group
  Grade 3 Drowsiness (N=30, 0) | 0.0 | NA — Event was not assessed in this group
  Appetite lost (N=30, 0) | 26.7 | NA — Event was not assessed in this group
  Grade 3 Appetite lost | 0.0 | NA — Event was not assessed in this group
  Irritability (N=30, 0) | 53.3 | NA — Event was not assessed in this group
  Grade 3 Irritability (N=30, 0) | 0.0 | NA — Event was not assessed in this group
  Headache (N=0, 30) | NA — Event was not assessed in this group | 10.0
  Grade 3 Headache (N=0, 30) | NA — Event was not assessed in this group | 0.0
  Malaise (N=0, 30) | NA — Event was not assessed in this group | 13.3
  Grade 3 Malaise (N=0, 30) | NA — Event was not assessed in this group | 0.0
  Myalgia (N=0, 30) | NA — Event was not assessed in this group | 13.3
  Grade 3 Myalgia (N=0, 30) | NA — Event was not assessed in this group | 0.0

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Antibodies Before and Post Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Geometric titers of influenza antibodies were assessed using the hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-final vaccination
Population: Geometric mean titers were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Number analyzed (Participants) | 29 | 29
Titers (1/dilutions)
  A/H1N1; Pre-vaccination | 32.6 [16.4 to 64.9] | 361 [179 to 727]
  A/H1N1; Post-vaccination | 447 [254 to 787] | 1235 [793 to 1924]
  A/H3N2; Pre-vaccination | 55.9 [25.7 to 121] | 277 [162 to 473]
  A/H3N2; Post-vaccination | 696 [416 to 1165] | 1250 [861 to 1814]
  B (Yamagata); Pre-vaccination | 56.6 [30.3 to 106] | 281 [158 to 497]
  B (Yamagata); Post-vaccination | 617 [342 to 1115] | 1425 [972 to 2090]
  B (Victoria); Pre-vaccination | 12.5 [6.88 to 22.9] | 156 [85.9 to 284]
  B (Victoria); Post-vaccination | 352 [203 to 612] | 1136 [706 to 1828]

3. Secondary Outcome: Number of Participants With Seroprotection Before and Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent Vaccine
Description: Influenza antibodies were assessed using the hemagglutination inhibition (HAI) assay. Seroprotection was defined as a titer ≥ 40 (l/dil) at pre-vaccination and at 28 days after the final vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-final vaccination
Population: Seroprotection was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Number analyzed (Participants) | 29 | 29
Percentage of participants
  A/H1N1; Pre-vaccination | 44.8 | 86.2
  A/H1N1; Post-vaccination | 93.1 | 96.6
  A/H3N2; Pre-vaccination | 62.1 | 93.1
  A/H3N2; Post-vaccination | 96.6 | 100.0
  B (Yamagata); Pre-vaccination | 55.2 | 89.7
  B (Yamagata); Post-vaccination | 100.0 | 100.0
  B (Victoria); Pre-vaccination | 17.2 | 82.8
  B (Victoria); Post-vaccination | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants With Seroconversion Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent Vaccine
Description: Influenza antibodies were assessed using the hemagglutination inhibition (HAI) assay. Seroconversion is defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 28 post-final vaccination
Population: Seroconversion was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Number analyzed (Participants) | 29 | 29
Percentage of participants
  A/H1N1 | 86.2 | 34.5
  A/H3N2 | 89.7 | 58.6
  B (Yamagata) | 86.2 | 58.6
  B (Victoria) | 89.7 | 69.0

5. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Influenza Antibodies Following Vaccination With the 2014-2015 Formulation of Fluzone® Quadrivalent Vaccine
Description: Geometric titer ratios of influenza antibodies were assessed using the hemagglutination inhibition (HAI) assay.
Time Frame: Day 28 post-final vaccination
Population: Geometric mean titer ratios were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Number analyzed (Participants) | 29 | 29
Titer ratio
  A/H1N1 | 10.9 [6.61 to 18.0] | 3.30 [2.14 to 5.11]
  A/H3N2 | 10.4 [6.59 to 16.4] | 4.51 [3.09 to 6.58]
  B (Yamagata) | 10.0 [6.35 to 15.9] | 5.02 [3.43 to 7.34]
  B (Victoria) | 18.9 [11.6 to 30.8] | 7.10 [4.71 to 10.7]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 7 post-any vaccination.
Arm/Group | 6 to < 36 Months of Age | 3 to < 9 Years of Age
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 21/30 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 to < 36 Months of Age (N=30) | 3 to < 9 Years of Age (N=30)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 6 to < 36 Months of Age (N=30) | 3 to < 9 Years of Age (N=30)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Injection site Tenderness (General disorders) | 21 (21) | 0 (0)
Injection site Erythema (General disorders) | 15 (15) | 20 (20)
Injection site Swelling (General disorders) | 7 (7) | 13 (13)
Fever (General disorders) | 6/29 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Crying abnormal (Psychiatric disorders) | 10 (10) | 0 (0)
Drowsiness (Nervous system disorders) | 9 (9) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 8 (8) | 0 (0)
Irritability (Psychiatric disorders) | 16 (16) | 0 (0)
Injection site Pain (General disorders) | 0 (0) | 22 (22)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications